CLINICAL TRIAL: NCT05534490
Title: The Investigation of the Effect of Foot Massage on the Functionality of Older Adults After General Surgery
Brief Title: Surgery and Functionality in Older Adults
Acronym: SFO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, asuman saltan, Associate Proffesor, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAD001
Record Dates: First submitted 2022-09-04; First posted 2022-09-09 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Fear; Movement Disorder, Functional; Kinesiophobia; Surgery
MeSH Terms: conditions — Conversion Disorder; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study, single-blind.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): The group will have a foot massage.
  Interventions: Other: therapatic Foot massaje (sweden technic)
- Control group (No Intervention): The group will not have any intervention.

INTERVENTIONS:
Other: therapatic Foot massaje (sweden technic) — Everything is explained to the individuals on the day of surgery. After the surgery, when the individuals regains consciousness in the service, the Swedish massage technique is applied bilaterally for 10 minutes. In addition to the demographic data of the patient before the application and in the preoperative period; pain, mental level, delirium status, mobility, kinesiophobia, balance, and functional independence level measurement evaluations are made. Massage is continued for a total of 20 minutes, 10 minutes for each foot, once a day until the patient is discharged. The measurements are repeated on the day the individual will be discharged.
  Arms: Massage group

SUMMARY:
When the literature is examined, it has not been found that the use of massage applications in relation to the functional level of individuals who have undergone abdominal surgery. We think that our study will be the first in this field. Therefore, this study will lay the groundwork for future studies on the subject. In the future, it is aimed to establish a standardized evaluation method to determine the functional levels of individuals who have undergone abdominal surgery and to determine the ideal duration and frequency when a decision is made to apply foot massage in the future with the data obtained as a result of this method. In this study, the effectiveness of foot massage on the functional level of individuals with high post-surgical kinesiophobia will be investigated.

DETAILED DESCRIPTION:
Pain, delirium, kinesiophobia, balance, mental level, and mobility are factors that express functional level in elderly individuals. It is especially important to regain at least the previous functional level after surgery. Although there are protocols and evaluation methods for returning or regaining the functional level after certain surgeries (for examples orthopedic surgeries such as knee or hip and cardiovascular surgery), admission to the discharge or rehabilitation program, especially after abdominal surgeries within the scope of general surgery. There is no protocol or evaluation method in the literature for the evaluation of situations such as In the studies, it was seen that scales were developed to evaluate the morbidity rate rather than the functional level after general surgery. Therefore, the evaluation of the functional level after surgery will be one of the important steps taken for the discharge or rehabilitation process to start as soon as possible. However, with the applications to reduce the high rate of kinesiophobia, the duration of discharge can be shortened, and rehabilitation can be started more quickly if necessary. With this study, the functional levels of the patients hospitalized in the general surgery service will be evaluated and the effect of foot massage on the functional level will be investigated. With this study, the effectiveness of foot massage on the functional level will be investigated in individuals with high post-surgical kinesiophobia, which is expected to be the first in the literature.

Our hypothesis (H0) is that foot massage after surgery has no effect on the functional level. Our H1 hypothesis is that foot massage has an effect on the functional level.

In light of the above information, in this study, a foot massage (Swedish massage) lasting 20 minutes in total, will be applied to the feet of the patients in the post-surgical service once a day, bilaterally, until discharge. Pain, mental level, delirium status, mobility, kinesiophobia, balance, and functional independence level measurements of the individual will be repeated before and after the massage.

The aim of this study is to investigate the effect of massage on the functional level of elderly individuals in the postoperative period. The study will be carried out between July 2022 and October 2022 in a randomized controlled manner in individuals aged 65-75 years in Kocaeli University Research and Practice Hospital general surgery clinic.

ELIGIBILITY:
Inclusion Criteria:

Lying in the service after surgery

Being in the age range of 65-75 years -

Exclusion Criteria:

Using sedative or narcotic drugs

Having vascular problems such as deep vein thrombosis in the feet

Having skin diseases such as ulcers, infections, fungi on the feet

Fracture of lower extremity

-

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Decreased Kinesiophobia | 3 weeks
  Measures will doing with Tampa scale of kinesiophobia.

SECONDARY OUTCOMES:
Decreased Pain | 3 weeks
  Measures will doing with Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: asuman saltan, Principal Investigator — YU
Locations (1):
- Asuman Saltan, Merkez, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saltan A, Mert S, Topbas O, Aksu B. The investigation of effect on foot plantar massage on functional recovery in older adults with general surgery, randomized clinical trial. Aging Clin Exp Res. 2024 May 23;36(1):118. doi: 10.1007/s40520-024-02770-2. PMID 38780814